CLINICAL TRIAL: NCT02975089
Title: A Pilot Study Comparing Effects of Nutrients Supplements and Dietary Approach in Frailty Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); Miao-Li General Hospital, Miao-Li City, Taiwan (Unknown)
Responsible Party: Principal Investigator, Wen-Harn Pan, Professor, Academia Sinica, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AS-IRB-BM-14044
Record Dates: First submitted 2016-09-21; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Frail Elderly
Keywords: Frailty; nutrition education; designed dishware; balanced diet; multiple dietary components
MeSH Terms: conditions — Frailty | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): A leaflet of healthy diet for elderly
- Nutritional Intervention 1 (Experimental): "Multi-nutrient" supplement
  Interventions: Dietary Supplement: "multi-nutrient" supplement
- Nutritional Intervention 2 (Experimental): "Multi-nutrient & soy protein" supplement
  Interventions: Dietary Supplement: "multi-nutrient & soy protein" supplement
- Nutritional Intervention 3 (Experimental): Nutrition education on balanced diet & food supplement
  Interventions: Dietary Supplement: Nutrition education on balanced diet & food supplement

INTERVENTIONS:
Dietary Supplement: "multi-nutrient" supplement — 1. 1.3g/d multivitamins & minerals powder
  2. Leaflet content (same as control)
  Arms: Nutritional Intervention 1
Dietary Supplement: "multi-nutrient & soy protein" supplement — 1. 1.3g/d multivitamins & minerals powder
  2. 16g/d isolated soy protein powder
  3. Leaflet content (same as control)
  Arms: Nutritional Intervention 2
Dietary Supplement: Nutrition education on balanced diet & food supplement — 1. Nutrition education with a designed plate
  2. 10g/d mixed nuts (cashews, pumpkin seeds, walnuts, macadamia, pine nuts, and almonds)
  3. 25g/d milk powder (skimmed and calcium added)
  4. Leaflet content (same as control)
  Arms: Nutritional Intervention 3

SUMMARY:
The proportion of the elderly population has increased rapidly worldwide. Frailty is a common geriatric syndrome. Comprehensive dietary management strategy may have beneficial effects on frailty prevention and reversal. We compared the effects between micronutrients and/or protein supplement, and balanced diet on frailty status in elderly individuals who were at either pre-frail or frail stage. A total of 37 subjects completed a 3-month paralleled, single-blind, randomized control trial on (1) multiple nutrients supplementations, (2) multiple nutrients plus isolated soy protein supplementation, and (3) individualized nutrition education with designed dishware for balanced diet as well as food supplementations (mixed nuts and milk powder). Intervention effects on dietary intakes, biomarkers, frailty score and geriatric depression score (GDS) were assessed. The nutrition education intervention with designed dishware and milk powder/nuts supplement significantly increased the intake of vegetables, dairy, and nuts, along with increased concentration of urinary urea nitrogen of the pre-frail/frail elders. It yielded a significant reduction in frailty score (p<0.05) and a borderline decrease (p=0.063) in GDS-SF. Our study indicated that the dietary approach with easy-to-comprehend dishware and food supplements to optimize the distribution of multiple dietary components showed its potential to improve not only frail status but also psychological condition in elderly.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years of age
* Have at least one of the modified Fried's Frailty phenotypes
* Sign informed consent form for study participation

Modified Fried's Frailty phenotypes:

1. unintentional weight loss > 5% or 3 kg in previous year
2. Exhaustion: defined as positive answer to the question "I had felt fatigue or exhaustion for >3 days in the previous week"
3. Weakness: hand grip strength is below the gender and BMI specific thresholds. The cutoff points are set as follows:

   Men: For BMI ≤ 22.1, < 25.0 kg; for BMI 22.1-24.3, < 26.5 kg; for BMI 24.4-26.3, < 26.4 kg; for BMI ≥ 26.3, < 27.2 kg Women: for BMI ≤ 22.3, <14.6 kg; for BMI 22.3-24.2, <16.1 kg; for BMI 24.3-26.8, <16.5 kg; for BMI ≥ 26.8, < 16.4 kg
4. Slowness: gait speed is slower than the gender and height specific thresholds. The cutoff points are set as follows:

   Men: for height ≤ 163 cm, >14.92 sec/10m; for > 163 cm, >=14.08 sec/10m Women: for height ≤ 152 cm, >17.54 sec/10m; for > 152 cm, >=14.92 sec/10m
5. Low Physical Activity: No exercise and no labor or leisure-time physical activity in the past year, or below the calorie consumption: men <594kcal/week and women <295kcal/week.

Exclusion Criteria:

1. Severe illness (such as cancer under treatment), being bed-ridden, or unable to move
2. Diagnosed dementia, depression, psychosis, mental disorder, or cannot be effectively communicated with（e.g., MMSE<16）
3. Dumbness, severe hearing or visual impairment, or unable to complete the interview
4. Institutionalized individuals, such as living in a long-term care facility or being hospitalized

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changed dietary intake | Change from Baseline to month 1 and to month 3
  Usual dietary intake was assessed by inquiring about most frequently consumed breakfast, lunch, dinner, and snack items and the corresponding amounts by licensed dietitians with the assistance of food models and measuring dishware. Dietary intake data were transformed into nutrient data, using a computerized worksheet based on Nutrition and Health Survey Food and Nutrient Database.

SECONDARY OUTCOMES:
Changed frailty score | Change from baseline to month 1 and to month 3
  All participants were evaluated for frailty, based on the modified Fried criteria. Five frail phenotypes were assigned: (1) unintentional weight loss, (2) self-reported exhaustion, (3) weak grip strength, (4) slow gait speed, and (5) low level of physical activity. For estimating frailty score, participants scored one point from each phenotype if any of which was satisfied with a maximal score of 5 in total. Participants were classified as pre-frail by one point, and as frail by 3 or more points, otherwise as robust.
Changed GDS-SF score | Change from Baseline to month 1 and to month 3
  Geriatric depression scale-short form (GDS-SF) Chinese version is a 15-item assessment used to identify depression in the elderly. Participants with 5-9 points were at risk of depression, and ≥10 points were depression.
Changed urinary urea nitrogen levels | Change from baseline to month 3
  The first morning urine sample was collected by subjects and brought into the hospital for analyzing urinary urea nitrogen.
Changed urine creatinine levels | Change from baseline to month 3
  The first morning urine sample was collected by subjects and brought into the hospital for analyzing urine creatinine.
Changed nutritional status | Change from Baseline to month 1 and to month 3
  Nutritional status was assessed by mini nutritional assessment-short form (MNA-SF). MNA-SF point ≥12 was of normal nutritional status; between 8 and 11 was at risk for malnutrition; ≤7 was at malnutrition status.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D., Principal Investigator — Institute of Biomedical Sciences, Academia Sinica